CLINICAL TRIAL: NCT01266837
Title: An Open Label, Single Arm Trial to Characterize Patients With Metastatic Renal Cell Carcinoma Treated With Everolimus After Failure of the First VEGF-targeted Therapy
Brief Title: Open Label, Single Arm Trial to Characterize Patients With Metastatic RCC Treated With Everolimus After Failure of the First VEGF-targeted Therapy (MARC-2)
Acronym: MARC-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: iOMEDICO AG (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001LDE36T; 2010-021370-11 (EudraCT Number)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Metastatic Renal Cell Carcinoma; Failure of Exactly One Prior VEGF-targeted Therapy
Keywords: metastatic renal cell carcinoma; biomarker; Everolimus
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Other): Treatment with Everolimus
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — 10 mg p.o once daily
  Other Names: Afinitor

SUMMARY:
A single arm, open-label, multi-center phase IV clinical trial for patients with metastatic renal cell carcinoma, who have progressed on or after the first VEGF-targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Aged 18 years and above
3. Histologically or cytologically confirmed predominantly clear cell renal cell carcinoma
4. Metastatic disease documented by CT or MRI (histological confirmation not mandatory but wishful)
5. Patients with or without nephrectomy (partial or total)
6. Patients with at least one measurable lesion at baseline according to RECIST criteria 1.1
7. Failure of exactly one prior VEGFR-TKI therapy (e.g. sunitinib, sorafenib, pazopanib) for metastatic renal cell carcinoma
8. ECOG 0-2
9. Hemoglobin ≥ 9.0 g/dL
10. Platelet count ≥75,000/μL
11. Absolute neutrophil count ≥1,5x109/l
12. Serum creatinine < 2.5 x ULN
13. Liver function: Serum bilirubin ≤ 1.5 x ULN, AST or ALT ≤ 2.5 x ULN. Patients with suspected liver metastasis: AST and ALT ≤ 5x ULN
14. Able to swallow the study drug whole as a tablet
15. Expected life expectancy of at least 6 months
16. Women of childbearing potential must have had a negative serum pregnancy test within 14 days prior to the administration of the study treatment or must have a documented condition that prohibits pregnancy (e.g. hysterectomy, post-menopausal).

Exclusion Criteria:

1. Patients who have received >1 prior VEGFR-TKI therapy or prior therapy with bevacizumab +/- interferon.
2. VEGFR-TKI therapy within 14 days prior to start of study drug
3. Patients who have previously received systemic mTOR inhibitors (sirolimus, temsirolimus, everolimus).
4. Patients with a known hypersensitivity to everolimus or other rapamycin (sirolimus, temsirolimus) or to its excipients.
5. Any condition which, in the opinion of the investigator, would preclude participation in this trial
6. Patients within 4 weeks post-major surgery (e.g., intra-thoracic, intra-abdominal or intrapelvic), open biopsy, or significant traumatic injury to avoid wound healing complications. Minor procedures and percutaneous biopsies or placement of vascular access device require 7 days prior to study entry.
7. Patients who had radiation therapy within 4 weeks prior to start of study treatment. Palliative radiotherapy to bone lesions within 2 weeks prior to study treatment start.
8. Patients in anticipation of the need for major surgical procedure during the course of the study.
9. Patients with a serious non-healing wound, ulcer, or bone fracture.
10. Patients with a history of seizure(s) not controlled with standard medical therapy.
11. History or clinical evidence of central nervous system (CNS) metastases. Subjects who have previously-treated CNS metastases (surgery ± radiotherapy, radiosurgery, or gamma knife) and meet all 3 of the following criteria are eligible:

    1. are asymptomatic and,
    2. have had no evidence of active CNS metastases for ≥ 3 months prior to enrolment (inactive/controlled CNS metastases are allowed) and,
    3. have no requirement for steroids or enzyme-inducing anticonvulsants (e.g. carbamazepine, phenobarbital, phenytoin)
12. Patients receiving chronic systemic treatment with corticosteroids (dose of > 10 mg/day methylprednisone equivalent) or another immunosuppressive agent. Inhaled and topical steroids are acceptable.
13. Poorly controlled diabetes as defined by fasting serum glucose >2.0 x ULN.
14. Impaired liver function classified as Child-Pugh class C.
15. Active (acute or chronic) or uncontrolled infection of bacterial, mycotic or viral genesis.
16. Liver disease such as chronic active hepatitis or chronic persistent hepatitis.
17. Patients with a known history of HIV seropositivity.
18. Patients with active bleeding disorders.
19. Patients who have any severe and/or uncontrolled medical conditions or other conditions within the past 12 months that could affect their participation in the study such as cardiac angioplasty or stenting, unstable angina pectoris, symptomatic peripheral vascular disease, symptomatic congestive heart failure (NYHA II, III, IV), myocardial infarction ≤ 6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia, any disorders that impair the ability to evaluate the patient or for the patient to complete the study.
20. Patients who have a history of another primary malignancy and off treatment for ≤ 3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of the uterine cervix or breast, and localized cancer of the bladder (T1) and prostate (T1 - T2).
21. Female patients who are pregnant or breast feeding.
22. Men and women of reproductive potential who are not using highly effective birth control methods. Oral contraceptives for female patients and barrier contraceptives are not acceptable. For definition of highly effective birth control methods please refer to section 12.3.6 of this protocol.
23. Patients who are using other investigational agents or who had received investigational drugs ≤ 2 weeks prior to study treatment start.
24. Patients unwilling or unable to comply with the protocol.
25. Exclusion criteria for MRI: intracorporal metal (e.g. incompatible heart valves, pacemakers), contrast media allergy, claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-03; Primary Completion 2017-09-26 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of patients progression free 6 months after start of study treatment | 2 years after LPI

SECONDARY OUTCOMES:
Relation between biomarkers and clinical benefit (response, stable disease and progression/ no clinical benefit) of patients | 2 years after LPI

CONTACTS AND LOCATIONS:
Overall Officials: Michael Staehler, Dr. med, Study Director — Ludwig-Maximilians-University Munich, Hospital Grosshadern
Locations (8):
- Germany (8):
  - Charitè Campus Benjamin Franklin, Berlin
  - Klinik und Poliklinik für Urologie , Universitätsklinikum Carl Gustav Carus der Technischen Universität Dresden, Dresden
  - Urologie - Waldkrankenhaus St. Marien, Erlangen
  - Klinik für Innere Medizin (Tumorforschung), Universitätsklinikum Essen, Essen
  - Zentrum Innere Medizin, Medizinische Hochschule Hannover, Hanover
  - Klinik für Urologie und Kinderurologie, Universitätsklinikum des Saarlandes, Homburg
  - Klinik für Urologie, Universitätsklinikum Jena, Jena
  - 5. Medizinische Klinik, Klinikum Nürnberg, Nuremberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staehler M, Stockle M, Christoph DC, Stenzl A, Potthoff K, Grimm MO, Klein D, Harde J, Bruning F, Goebell PJ, Augustin M, Roos F, Benz-Rud I, Marschner N, Grunwald V. Everolimus after failure of one prior VEGF-targeted therapy in metastatic renal cell carcinoma: Final results of the MARC-2 trial. Int J Cancer. 2021 Apr 1;148(7):1685-1694. doi: 10.1002/ijc.33349. Epub 2020 Oct 26. PMID 33070307